CLINICAL TRIAL: NCT03537495
Title: Short Intervention and Measurement of Pharmacokinetics of Linezolid in Tuberculosis Meningitis: a Pharmacokinetics and Safety/Tolerability Study
Brief Title: Pharmacokinetic Study of Linezolid for TB Meningitis
Acronym: SIMPLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Collaborators: Radboud University Medical Center (Other); Global Alliance for TB Drug Development (Other)
Responsible Party: Principal Investigator, Ahmad Rizal Ganiem, MD, PhD, Universitas Padjadjaran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TB-201805.01
Record Dates: First submitted 2018-05-02; First posted 2018-05-25 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Tuberculosis, Meningeal; Linezolid
Keywords: tuberculous meningitis; linezolid; pharmacokinetic study
MeSH Terms: conditions — Tuberculosis, Meningeal | interventions — Linezolid

STUDY DESIGN:
Intervention Model Description: TB meningitis patients will be randomised into three treatment groups to either receive no linezolid (control group); or 600 mg QD or 1200 mg QD linezolid next to high dose rifampicin (~35 mg/kg, based on weight), isoniazid (H) 300 mg, pyrazinamide (Z) 1500 mg and ethambutol (E) 750 mg once daily administered orally for 14 days. All patients will receive dexamethasone according to standard dosing in TBM.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm (No Intervention): Subjects in this arm will only receive high-dose rifampicin (~35 mg/kg, based on weight), isoniazid (H) 300 mg, pyrazinamide (Z) 1500 mg and ethambutol (E) 750 mg once daily administered orally for 14 days.
  High-dose rifampicin will consist of weight-banded fixed-dose combination (FDC), including rifampicin (R), isoniazid (H), pyrazinamide (Z) and ethambutol (E) according to international guidelines, combined with 900 mg rifampicin (≤37 kg: two 450 mg tablets) or 1200 mg rifampicin (>37 kg: two 600 mg tablets) to reach ~35 mg/kg rifampicin in total.
- Linezolid 600 (Experimental): Subjects in this arm will receive 600 mg linezolid QD along with high-dose rifampicin (~35 mg/kg, based on weight), isoniazid (H) 300 mg, pyrazinamide (Z) 1500 mg and ethambutol (E) 750 mg once daily administered orally for 14 days.
  Interventions: Drug: Linezolid
- Linezolid 1200 (Experimental): Subjects in this arm will receive 1200 mg linezolid QD along with rifampicin 1350 mg (~35 mg/kg, based on weight), isoniazid (H) 300 mg, pyrazinamide (Z) 1500 mg and ethambutol (E) 750 mg once daily administered orally for 14 days.
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Linezolid — Overall, there is an urgent need for improvement of TBM treatment. LInezolid is known to be well-penetrated to blood brain barrier. A combination of high-dose rifampicin and linezolid as an intensified add-on therapy in the management of TB meningitis has never been studied.
  The goal is to assess the most appropriate dose of linezolid for larger follow-up studies and to evaluate the feasibility of a linezolid-containing TBM regimen.
  Arms: Linezolid 1200; Linezolid 600

SUMMARY:
Tuberculosis meningitis (TBM) is the most severe manifestation of TB, resulting in death or neurological disability in up to 50% of affected patients, despite antibacterial treatment. This TBM treatment follows the model for pulmonary TB by using the same first-line TB drugs (a combination of rifampicin, isoniazid, pyrazinamide and ethambutol) and the same dosing guidelines, although it is known that penetration of two of these drugs (rifampicin and ethambutol) into cerebrospinal fluid (CSF) is limited. Improvement of treatment of TBM is urgently needed.

To do so, a combination of two interventions will be investigated in this study. A series of phase II clinical trials on higher doses of the pivotal TB drug rifampicin in Indonesian patients with TBM have shown that the dose of rifampicin can be increased from 10 mg/kg orally (standard dose) up to 30 mg/kg orally, resulting in a strong increase in exposure to this drug in plasma and CSF, no increase in grade III or IV adverse effects, and a reduction in mortality. Similarly, higher doses of rifampicin up to 35 mg/kg resulted in strong increases in plasma concentrations; the doses were well tolerated and reduced time to sputum conversion in African pulmonary TB patients.

Next to a higher dose of rifampicin, the approved antibacterial drug linezolid seems a good candidate for a new TBM regimen. The drug penetrates well into the CSF and is applied successfully against other central nervous system (CNS) infections (e.g. caused by penicillin-nonsusceptible Streptococcus pneumoniae, vancomycin-resistant enterococci and methicillin-resistant Staphylococcus aureus). In a study in China, linezolid in a dose of 600 mg BID orally strongly increased recovery of patients with TBM response. Linezolid is also being investigated as a new drug for (drug-resistant) pulmonary TB in numerous studies, in a dose of 1200 mg once daily. More severe adverse effects to this drug typically occur only after prolonged treatment during several months, not during short-term treatment.

Overall, linezolid is expected to be a promising and tolerable candidate for a new intensified TBM treatment regimen consisting of a backbone of high dose rifampicin plus linezolid.

DETAILED DESCRIPTION:
Overall aim is to determine the most appropriate dose of linezolid in the treatment of TB meningitis, when combined with high-dose rifampicin (35 mg/kg orally), to be tested in larger clinical follow-up studies.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years old or older
* Clinically diagnosed as TB meningitis patient
* CSF/blood glucose ratio < 0.5
* Willing to participate in the study by signing informed consent

Exclusion Criteria:

Patients who have one of the following criteria will be excluded:

* Failure to diagnostic lumbar puncture
* Confirmed cryptococcus meningitis (LFA) in HIV-positive patients; or diagnosed as bacterial meningitis based on clinical assessment and routine CSF examination.
* Treatment for tuberculosis for more than 3 days before admission
* History of TBM
* Current treatment with: MAO inhibitors, direct and indirect acting sympathomimetic drugs, vasopressive drugs, dopaminergic compounds, buspiron, serotonin reuptake inhibitors, tricyclic antidepressants, triptans, tramadol and meperidine
* History (< 2 weeks before start of linezolid) of taking any MAO inhibitors
* Pregnant or lactating females
* Hepatic insufficiency (ALT>5x upper normal limit)
* Kidney dysfunction (eGFR <50ml/min)
* Known hypersensitivity to rifampicin and/or linezolid
* Rapid clinical deterioration at time of presentation (sepsis, decreasing consciousness, or signs of cerebral oedema or herniation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Linezolid exposure in blood and CSF | day 2 and day 11
  Linezolid exposure in blood (full plasma concentration-versus-time profiles (0-24h)) will be measured in 2 days, i.e. day 2 (+/- 1) and at day 11 (+/- 1) of TB treatment. In each sampling day, there will be 6 sampling points i.e. at 0 (pre-dose), 1, 2, 4, 8, and 12 h after study medication intake
  One CSF sample per patient will be taken at the same day as PK sampling i.e. at 2, 4 or 8 hours post dose.

SECONDARY OUTCOMES:
Serious adverse event | Day 3, 7, 10 and 14
  Serious adverse events assessed daily during the 14 days of intensified treatment (e.g. gastro-intestinal intolerance), and grade 1-4 adverse events (e.g. liver function and hematology) assessed at day 3, 7, 10 and 14.
Clinical response | Day 3, 7 and 14.
  Clinical response includes resolution of fever, resolution of hyponatremia etc.
Neurological response | Day 3, 7 and 14.
  Neurological response includes resolution of consciousness, development of raised intracranial pressure, etc.
Mortality | Within 14 days and 1 month after starting treatment
  mortality during the first month will be recorded and cause of death will be classified as neurologic or non-neurologic, if applicable
Blood inflammatory response | at PK days (day 2 and 11), and day 7 and 14
  Profile of inflammatory response in blood
CSF inflammatory response | at PK sampling days (day 2 and 11)
  inflammatory response in CSF at PK sampling days

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad R Ganiem, MD, PhD, Principal Investigator — Hasan Sadikin General Hospital, Bandung, Indonesia
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruslami R, Ganiem AR, Dian S, Apriani L, Achmad TH, van der Ven AJ, Borm G, Aarnoutse RE, van Crevel R. Intensified regimen containing rifampicin and moxifloxacin for tuberculous meningitis: an open-label, randomised controlled phase 2 trial. Lancet Infect Dis. 2013 Jan;13(1):27-35. doi: 10.1016/S1473-3099(12)70264-5. Epub 2012 Oct 25. PMID 23103177
- [Background] Dian S, Yunivita V, Ganiem AR, Pramaesya T, Chaidir L, Wahyudi K, Achmad TH, Colbers A, Te Brake L, van Crevel R, Ruslami R, Aarnoutse R. Double-Blind, Randomized, Placebo-Controlled Phase II Dose-Finding Study To Evaluate High-Dose Rifampin for Tuberculous Meningitis. Antimicrob Agents Chemother. 2018 Nov 26;62(12):e01014-18. doi: 10.1128/AAC.01014-18. Print 2018 Dec. PMID 30224533